CLINICAL TRIAL: NCT04193969
Title: The Association Between Changes in Radicular Pain and Pain Modulation Among Patients With Lumbar Radiculopathy: A Pilot Study.
Brief Title: Changes in Radicular Pain and Pain Modulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spine Centre of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: S-20190091
Record Dates: First submitted 2019-11-24; First posted 2019-12-11 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Back Pain; Back Pain With Radiation
Keywords: low back pain; radiculopathy; conditioned pain modulation; temporal summation
MeSH Terms: conditions — Back Pain; Low Back Pain; Radiculopathy | interventions — Postsynaptic Potential Summation; Pain Measurement; Disability Evaluation

STUDY DESIGN:
Intervention Model Description: The study has a cohort design and will include a patient group (male and female) attending a treatment program at the Spine Centre of Southern Denmark and an equally large control group matched on age and gender.
Who Masked: Participant
Masking Description: The participants are not informed about test results during or after the sessions. The test equipment is computer controlled and user independent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiculopathy due to nerve root compression (Experimental): Participants with radicular leg pain due to lumbar disc herniation or to foraminal- or recess stenosis.
  Baseline assessments of pain intensities are performed through questionnaires prior to protocol. Data regarding initial pain, function, age, gender, pain-duration, weight and height is retrieved from the clinical registry SpineData.
  Pain sensitivity, temporal summation and conditioned pain modulation are assessed at the first visit in the treatment program. The protocol is repeated at the last visit in the treatment program.
  Interventions: Diagnostic Test: Pressure pain assessment using computer controlled cuff algometry; Diagnostic Test: Temporal summation (TS); Diagnostic Test: Conditioned pain modulation (CPM); Diagnostic Test: Low back pain rating scale (LBPRS-pain); Diagnostic Test: Oswestry Disability Index
- Healthy controls (Experimental): Healthy controls Healthy age and gender-matched controls. Gender, weight and height are registered on questionnaires prior to protocol.
  Pain sensitivity, temporal summation and conditioned pain modulation are assessed at the first visit. The tests are repeated at the next visit. The interval between the two sessions will be determined by the averaged interval between tests in the patient group.
  Interventions: Diagnostic Test: Pressure pain assessment using computer controlled cuff algometry; Diagnostic Test: Temporal summation (TS); Diagnostic Test: Conditioned pain modulation (CPM)

INTERVENTIONS:
Diagnostic Test: Pressure pain assessment using computer controlled cuff algometry — Pressure pain sensitivity is assessed. The pressure is gradually increased and pain is rated by the participant on an electronic visual analogue pain rating scale (VAS) which is connected to the equipment. The assessment is performed on the lower leg and the upper arm. The pain free leg and the left upper arm is used in the patient group. The leg used in the control group will be chosen in a balanced manner meaning that half will receive pressure on the left leg and the other half on the right leg. The pain detection threshold (PDT), pain pressure tolerance threshold (PPT) and pressure pain intensity perceived as 6 on the VAS (VAS6) at the leg site is registered. The PDT and PPT on the arm site is registered.
  Other Names: Assessment of pain sensitivity
Diagnostic Test: Temporal summation (TS) — 10 repeated inflations on the lower leg with a 1 sec interval. The pressure used at each pressure is equivalent the PPT measured at baseline. Each inflation is rated on the VAS. TS is registered as the increase pain intensity.
  Other Names: Repeated pressure pain
Diagnostic Test: Conditioned pain modulation (CPM) — The cuff on the upper arm is inflated until 70% of the PPT is reached. While the pressure on the arm is kept constant the cuff on the leg is inflated. PDT, PPT and VAS6 pressure at the leg site is registered during the tonic stimulation (pressure on the left arm). The procedure on the leg is repeated within 30 seconds after the pressure is released on the arm site.
  Other Names: Pain inhibition
Diagnostic Test: Low back pain rating scale (LBPRS-pain) — A questionnaire measuring the intensities of low back pain and leg pain currently, on average the last two weeks and the worst pain within the same period.
  Other Names: Pain intensity
  Arms: Radiculopathy due to nerve root compression
Diagnostic Test: Oswestry Disability Index — A questionnaire measuring the disability in relation to low back pain and leg pain.
  Other Names: Disability
  Arms: Radiculopathy due to nerve root compression

SUMMARY:
The objectives of this study are: 1)To investigate the difference in pain modulatory mechanisms using quantitative sensory testing (QST) between healthy controls and patients with radicular leg pain due to nerve root compression. 2) To investigate the association between changes in radiating leg pain and pain modulation among the patient group.

DETAILED DESCRIPTION:
Few studies have investigated pain modulatory mechanisms using QST in patients with lumbar radiculopathy due to nerve root compression. Knowledge about the association between changes in the experience of pain and changes measures of pain modulation is to our knowledge limited. The results could potentially contribute to knowledge about mechanisms involved in lumbar radiculopathy and facilitate future studies. The hypotheses of the study are: 1) Measures of pain modulation will be less efficient among patients with lumbar radiculopathy showing reduced pain inhibition and facilitated temporal summation compared to healthy controls. 2) Improvements in pain modulation will be associated with improvements in clinical pain outcomes

ELIGIBILITY:
Inclusion Criteria:

Patient group

* Radiating leg pain due to nerve root compression verified by MRI
* Clinical findings in accordance with MRI findings
* Average leg pain ≥ 3/10 on a numeric pain rating scale Controls
* No current or previous history of ongoing musculoskeletal pain

Exclusion Criteria:

Applies for both groups.

* Other specific medical conditions e.g. rheumatologic disease, diabetes or vascular diseases.
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Cuff sensitivity, measured with computer-controlled cuff algometry | At baseline and at discharge from treatment throughout study completion, an average of 6 months. The timeframe between the baseline test and follow up test for controls will be matched the patient group.
  Change in pain sensitivity between baseline and follow-up. Cuff is placed around the lower leg and on the upper arm and gradually inflated (1kPa/sec) on each location separately. In patients, the cuff is placed on the non-painful leg and left upper arm, in healthy controls, half of the participants the cuff is placed on the left leg and half on the right leg, while the other cuff is placed on the left upper arm. First, the pressure needed to evoke an onset of pain (pain detection threshold, PDT), the pressure at pain intensity VAS 6 (Measured on an electronic visual analogue scale: 0=No pain, 10=worst pain imaginable pain) and pain tolerance threshold (PTT) is assessed on the lower leg. Secondly, the PDT and the PTT is assessed on the left upper arm.
Temporal summation of pain (increase in pain during repeated pain stimuli at same intensity) measured with computer-controlled cuff algometry | At baseline and at discharge from treatment throughout study completion, an average of 6 months. The timeframe between the baseline test and follow up test for controls will be matched the patient group.
  Change in pain intensity between baseline and follow-up. Cuff is placed on the lower leg. In patients the non-painful leg is used, in healthy controls, half of the participants will be tested on the left leg and half on the right leg. 10 painful stimuli are performed with a one-second interval in between. After each stimulus, the participant rates the pain intensities using an electronic VAS ( 0=No pain, 10=worst pain imaginable pain). The increase in pain intensity is defined as temporal summation.
Conditioned pain modulation (change in pain sensitivity during a competing pain stimulus) measured with computer-controlled cuff algometry | At baseline and at discharge from treatment throughout study completion, an average of 6 months. The timeframe between the baseline test and follow up test for controls will be matched the patient group.
  Change in pain intensity between baseline and follow-up. Cuff is placed on the lower leg. In patients the non-painful leg is used, in healthy controls, half of the participants will be tested on the left leg and half on the right leg. 10 painful stimuli are performed with a one-second interval in between. After each stimulus, the participant rates the pain intensities using an electronic VAS ( 0=No pain, 10=worst pain imaginable pain). The increase in pain intensity is defined as temporal summation.

SECONDARY OUTCOMES:
Leg pain (measured on the low back pain rating scale) | At baseline and at discharge from treatment throughout study completion, an average of 6 months.
  Change in pain between post-treatment and pre-treatment. The average pain during the last two weeks, the worst pain experienced during the same period and current pain is rated by the patient. Range 0-30. 0=no pain, 30= Worst pain imaginable.
Back pain and leg pain (measured on the low back pain rating scale) | At baseline and at discharge from treatment throughout study completion, an average of 6 months.
  Change in pain between post-treatment and pre-treatment. Low back pain rating scale (LBPRS - pain): Two questionnaires with three numeric 11-point box scales (0-10) regarding low back pain and leg pain respectively. The average pain during the last two weeks, the worst pain experienced during the same period and current pain is rated by the patient. Range 0-60. 0=no pain, 60= Worst pain imaginable.
Disability (Measured on the Oswestry Disability index) | At baseline and at discharge from treatment throughout study completion, an average of 6 months.
  Change in disability between post-treatment and pretreatment. Range 0-100, 0= No disability, 100 maximum disability possible.

CONTACTS AND LOCATIONS:
Overall Officials: Berit Schiøtzz-Christensen, Professor, Principal Investigator — Research department of Spine Center of Southern Denmark
Locations (1):
- Spine Centre of Southern Denmark, Middelfart, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaegter HB, Palsson TS, Graven-Nielsen T. Facilitated Pronociceptive Pain Mechanisms in Radiating Back Pain Compared With Localized Back Pain. J Pain. 2017 Aug;18(8):973-983. doi: 10.1016/j.jpain.2017.03.002. Epub 2017 Mar 24. PMID 28344100
- [Background] Mehta V, Snidvongs S, Ghai B, Langford R, Wodehouse T. Characterization of peripheral and central sensitization after dorsal root ganglion intervention in patients with unilateral lumbosacral radicular pain: a prospective pilot study. Br J Anaesth. 2017 Jun 1;118(6):924-931. doi: 10.1093/bja/aex089. PMID 28575334
- [Background] Yarnitsky D. Role of endogenous pain modulation in chronic pain mechanisms and treatment. Pain. 2015 Apr;156 Suppl 1:S24-S31. doi: 10.1097/01.j.pain.0000460343.46847.58. PMID 25789433
- [Background] Graven-Nielsen T, Izumi M, Petersen KK, Arendt-Nielsen L. User-independent assessment of conditioning pain modulation by cuff pressure algometry. Eur J Pain. 2017 Mar;21(3):552-561. doi: 10.1002/ejp.958. Epub 2016 Nov 11. PMID 27859944
- [Background] Graven-Nielsen T, Vaegter HB, Finocchietti S, Handberg G, Arendt-Nielsen L. Assessment of musculoskeletal pain sensitivity and temporal summation by cuff pressure algometry: a reliability study. Pain. 2015 Nov;156(11):2193-2202. doi: 10.1097/j.pain.0000000000000294. PMID 26172551